CLINICAL TRIAL: NCT05270642
Title: Research on Intelligent System of Plan for Microwave Thermal Field for Hepatocellular Carcinoma
Brief Title: Plan for Microwave Thermal Field
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, M.D., Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2021-439-01
Record Dates: First submitted 2022-02-27; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma; Ablation
Keywords: hepatocellular Carcinoma; microwave ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCC patients guided by Plan for Microwave Thermal Field (Experimental): The plan for HCC patients undergoing microwave ablation would be refer to Plan for Microwave Thermal Field system
  Interventions: Procedure: Microwave Thermal guided by Plan for Microwave Thermal Field system

INTERVENTIONS:
Procedure: Microwave Thermal guided by Plan for Microwave Thermal Field system — When HCC patients undergo microwave ablation, the doctor will refer to the ablation plan provided by the system.If the plan is consistent with what the doctor thinks, follow the plan provided by the system. If the protocol is not consistent with what the doctor thinks, the doctor will revise the protocol.

SUMMARY:
Develop an intelligent system based on contrast-enhanced ultrasound and clinical information to help doctors automatically obtain ablation parameters (ablation needle number, ablation needle type, ablation time,ablation power) when preparing to use microwave ablation to treat hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy or clinical diagnosis of HCC
2. Complete clinical information and preoperative CEUS
3. Curative treatment

Exclusion Criteria:

1. Palliative care
2. Intolerance to ablation
3. Severe coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
MRI within 3 days after ablation | MRI within 3 days after ablation
  Postoperative MRI is used to determine whether the ablation zone completely covers the tumor and whether the size is appropriate
local tumor progression | 6 months
  Follow up to observe whether local tumor progression occurs within 6 months after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided